CLINICAL TRIAL: NCT03379870
Title: Outcomes in Children With Cochlear Implants and Pre-Operative Residual Hearing: Electric Only and Electric-Acoustic Stimulation
Brief Title: Outcomes in Children With Pre-operative Residual Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-2360
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-05

CONDITIONS: High Frequency Sensorineural Hearing Impairment; Hearing Disorders in Children
Keywords: cochlear implant; electric acoustic stimulation; EAS; hearing loss; pediatric
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EAS Arm (Experimental): Subjects who receive a CI and present with a post-operative LFPTA of ≤ 75 dB HL.
  Electric Acoustic Speech Processor: Electric-acoustic stimulation (EAS) fitting.
  Interventions: Device: Electric Acoustic Speech Processor: Electric-acoustic stimulation fitting
- FES Arm (Experimental): Subjects with pre-operative low frequency hearing who receive a CI and present with a post-operative LFPTA of > 75 dB HL.
  Electric Acoustic Speech Processor: Full-electric stimulation (FES) fitting
  Interventions: Device: Electric Acoustic Speech Processor: Full-electric stimulation fitting

INTERVENTIONS:
Device: Electric Acoustic Speech Processor: Electric-acoustic stimulation fitting — Electric Acoustic Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or better,
  Other Names: MED-EL SONNET EAS; MED-EL SONNET 2 EAS
  Arms: EAS Arm
Device: Electric Acoustic Speech Processor: Full-electric stimulation fitting — Electric Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or poorer and pre-operative low frequency hearing averages of 75 dB HL or better.
  Other Names: MED-EL SONNET EAS; MED-EL SONNET 2 EAS
  Arms: FES Arm

SUMMARY:
Purpose: Routine clinical care and pilot study data has shown evidence of postoperative hearing preservation in pediatric cochlear implant (CI) recipients. The primary aim of this study is to investigate speech perception performance in pediatric CI recipients with functional pre-operative hearing.

Participants: Two cohorts of CI recipients aged 6 through 17 years who had pre-operative low frequency residual hearing. Subjects in Arm 1 (EAS Arm; electric-acoustic stimulation) will present with a post-operative low frequency pure tone average (125, 250, and 500 Hz) of ≤ 75 dB HL, and those in Arm 2 (FES Arm; full-electric stimulation) will present with a post-operative low frequency pure tone average (LFPTA) that exceeds 75 dB HL.

Procedures (methods): Subjects will complete speech perception and quality of life testing during post-operative intervals. Subjects in the EAS Arm will be evaluated with combined electric-acoustic stimulation (EAS). Subjects in FES Arm will be evaluated with FES alone.

DETAILED DESCRIPTION:
As children with more residual hearing are receiving cochlear implants (CIs), there is an opportunity to preserve that hearing and provide combined electric and acoustic stimulation (EAS). The primary aim of this study is to investigate speech perception performance in pediatric CI recipients with functional pre-operative hearing. Specifically, the investigators intend to compare speech understanding using EAS and traditional full electric stimulation.

While hearing preservation rates are good, they are not guaranteed. Children with progressive hearing loss may continue to lose hearing, even if they maintain some residual hearing immediately after surgery. As a secondary aim, the investigators intend to study outcomes in children who do not maintain residual hearing and are fit with traditional CI programming methods. Children with more residual hearing are being implanted, and this study design allows validation of outcomes in both populations.

Subject enrollment will occur on the initial stimulation date. Those who have maintained a low frequency hearing average of 75 dB HL or better will be fit with a SONNET EAS or SONNET 2 EAS device using combined acoustic and electric stimulation. Those who have not maintained low frequency hearing will be fit with a SONNET EAS or SONNET 2 EAS device using electric stimulation only. Subjects will be followed at regular intervals throughout the year duration of the study and will be tested on measures of speech understanding in quiet, speech understanding in noise, quality of life, and discrimination of prosody or pitch changes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 through 17 years
* Spoken English as the primary language (speech perception testing conducted in English).
* Recipient of a MED-EL SYNCHRONY Cochlear Implant device.
* Pre-operative LFPTA of ≤ 75 dB HL.
* Willing and able to participate in study procedures.
* Realistic parental/patient expectations.
* Language skills judged to be adequate enough to perform study tasks.

Exclusion Criteria:

* Inability to perform open set speech perception due to oral motor delays.
* Inability to perform test battery due to behavior or cognitive impairment
* Unwilling or unable to participate in study procedures.
* Cochlear nerve deficiency.
* Anatomical considerations that necessitated surgical modifications such as ossification, incomplete insertion, or placement in scala vestibuli.

Ages: 60 Months to 215 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Park, AuD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The Children's Cochlear Implant Center at UNC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EAS Arm: Subjects who receive a CI and present with a post-operative LFPTA of ≤ 75 dB HL.
  Electric Acoustic Speech Processor: EAS fitting.
  EAS fitting: Electric Acoustic Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or better,
- FES Arm: Subjects with pre-operative low frequency hearing who receive a CI and present with a post-operative LFPTA of > 75 dB HL.
  Electric Acoustic Speech Processor: FES fitting
  FES fitting: Full-electric stimulation for children with post-operative residual low frequency hearing averages greater than 75 dB HL and pre-operative low frequency hearing averages of 75 dB HL or better.
Period: Overall Study
Arm/Group | EAS Arm | FES Arm
Started | 16 | 12
Completed | 14 | 11
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- EAS Arm: Subjects who receive a CI and present with a post-operative LFPTA of ≤ 75 dB HL.
  Electric Acoustic Speech Processor: EAS fitting: Electric Acoustic Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or better.
- FES Arm: Subjects with pre-operative low frequency hearing who receive a CI and present with a post-operative LFPTA of > 75 dB HL.
  Electric Acoustic Speech Processor: Electric only fitting: Electric Stimulation for children with post-operative residual low frequency hearing averages greater than 75 dB HL and pre-operative low frequency hearing averages of 75 dB HL or better.
- Total: Total of all reporting groups
Arm/Group | EAS Arm | FES Arm | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (3.9) | 10.5 (3.3) | 10.2 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 25
Pre-operative Low Frequency Pure Tone Average (PTA) [Mean (Standard Deviation); unit: Decibels (dB)] — Average hearing levels measured in decibels (dB) as measured at 125, 250, and 500 Hz
  Decibels (dB) | 29.9 (17.8) | 57.5 (11.6) | 43.1 (20.5)
Post-operative Low Frequency Pure Tone Average (PTA) at Enrollment [Mean (Standard Deviation); unit: Decibels (dB)] — Average of thresholds measured at 125, 250, and 500 Hz at enrollment.
  Decibels (dB) | 46.2 (14.5) | 85.8 (16.4) | 63.6 (25.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean CNC Word Scores
Description: The Consonant Nucleus Consonant (CNC) word list is established as a standard test of speech perception outcomes. Results for EAS and FES Arms at 12 months post stimulation will be compared. Lower scores indicate a poorer outcome and higher scores a better outcome. Scale 0 - 100%
Time Frame: 12 months post stimulation
Population: Subjects who completed the 12-month protocol
Measure: Mean (Standard Deviation); unit: Percent Correct
Groups:
- EAS Arm: Subjects who receive a CI and present with a post-operative LFPTA of ≤ 75 dB HL.
  Electric Acoustic Speech Processor: EAS fitting: Electric Acoustic Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or better,
- FES Arm: Subjects with pre-operative low frequency hearing who receive a CI and present with a post-operative LFPTA of > 75 dB HL.
  Electric Acoustic Speech Processor: Electric only fitting: Electric Stimulation for children with post-operative residual low frequency hearing averages poorer than 75 dB HL and pre-operative low frequency hearing averages of 75 dB HL or better.
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 14 | 11
Percent Correct | 71.0 (18.0) | 68.4 (26.0)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed Consonant Nucleus Consonant (CNC) Word scores obtained 12-months post-activation to evaluate differences between groups. Percent correct data were converted to rationalized arcsine units (RAU) prior to data analysis to control for potential floor or ceiling effects (e.g., scores <20%); p = .768, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

2. Primary Outcome: Mean BKB-SIN SNR-50 Scores
Description: Sentences and babble will be presented from the same speaker. An average score known as the SNR-50 will be obtained in both conditions. The SNR-50 score is an estimate of the signal-to-noise ratio associated with 50% correct based on word-level scoring. Results for EAS and FES listeners at 12 months post stimulation will be compared. In this test, lower scores indicate a better outcome and higher scores a poorer outcome. Scores range from -6 dB to +21 dB.
Time Frame: 12 months post-stimulation
Population: Subjects who completed the 12-month protocol
Measure: Mean (Standard Deviation); unit: Signal to noise ratio (SNR) in decibels
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 14 | 11
Signal to noise ratio (SNR) in decibels | 6.9 (9.3) | 5.5 (7.7)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed BKB-SIN scores obtained 12-months post-activation to evaluate differences between groups. Scores range from -6 to +21 and lower scores are better; p = .529, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

3. Secondary Outcome: Mean Pediatric SSQ Scores
Description: The Speech, Spatial, and Qualities of Hearing (SSQ) Scale assesses performance in three domains, hearing speech in quiet and noise environments (9 items), spatial or directional hearing (5 items) and sound qualities (8 items), which address sound segregation and listening effort. Each item is rated on a 11-point scale, with 0 as the lowest possible performance and 10 as the highest. Domain scores represent an average of item ratings. There is a version for children that will be used for this study. Lower scores indicate a poorer outcome, and higher scores a better outcome.
Time Frame: Baseline, 12 months post-stimulation
Population: Subjects who completed the 12-month protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 14 | 11
score on a scale
  Pre-operative | 4.5 (2.3) | 4.4 (2.1)
  12-months post activation | 7.1 (2.1) | 6.7 (1.9)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed SSQ scores obtained pre-operatively and at 12-months post-activation to evaluate benefit of cochlear implantation; p = .010, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

4. Secondary Outcome: Receptive Language Scores
Description: Mean receptive language scores as measured by the Oral and Written Language Scales, 2nd edition (OWLS II), comparing pre-operative scores to the 12 month test point for both groups. These tests are normed and reported as scaled scores. T-Scores scores will be compared. Low scores are indicative of a poorer outcome, and higher scores a better outcome. A scores of 100 indicated the population mean with a standard deviation of 15. A score of 85 or poorer is indicative of a receptive language delay.
Time Frame: 12 months post-stimulation
Population: Not all participants were tested pre-operatively
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 13 | 10
T-score
  Pre-operatively: number analyzed (Participants) | 11 | 9
  Pre-operatively | 98.8 (19.5) | 99.8 (20.3)
  12-months post activation | 100.1 (16.2) | 89.7 (22.0)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed receptive language scores pre-operatively and 12-months post activation to test for change over time and differences between groups; p > .069, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05

5. Secondary Outcome: Articulation Scores
Description: Mean articulation scores as measured by the Goldman-Fristoe Test of Articulation, 3rd edition (GFTA3), comparing pre-operative scores to the 12 month test point for both groups. These tests are normed and reported as scaled scores. T-Scores scores will be compared. Low scores are indicative of a poorer outcome, and higher scores a better outcome. A score of 100 indicates the population mean with a standard deviation of 15. A score of 85 or poorer is indicative of a articulation delay.
Time Frame: 12 months post-stimulation
Population: Data reported for all subjects who completed pre-operative testing.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 12 | 10
T-score
  Pre-operative | 86.8 (14.4) | 83.6 (23.2)
  12-months post activation | 99.3 (20.1) | 88.3 (18.8)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed articulation scores pre-operative and 12-months post activation to test for change over time and differences between groups; p = .02, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05; Main effect of test point (pre-operative vs post-activation)

6. Secondary Outcome: Expressive Language Scores
Description: Mean expressive language scores as measured by the Oral and Written Language Scales, 2nd edition (OWLS II), comparing pre-operative scores to the 12 month test point for both groups. These tests are normed and reported as scaled scores. T-Scores scores will be compared. Low scores are indicative of a poorer outcome, and higher scores a better outcome. A score of 100 indicates the population mean with a standard deviation of 15. A score of 85 or poorer is indicative of an expressive language delay.
Time Frame: 12 months post-stimulation
Population: Not all subjects completed pre-operative testing
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EAS Arm | FES Arm
Number analyzed (Participants) | 13 | 10
T-score
  Pre-operative: number analyzed (Participants) | 11 | 9
  Pre-operative | 96.8 (17.2) | 99.7 (12.2)
  12-months post activation | 101.9 (18.0) | 97.6 (22.0)
Statistical Analysis 1: Comparison: EAS Arm vs FES Arm; Test type: Superiority — Analyzed expressive language scores pre-operatively and 12-months post activation to test for change over time and differences between groups; p = .007, Mixed Models Analysis — The a priori threshold for statistical significance was < 0.05; Main effect of test point (pre-operative vs post activation)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through 12 months post-activation.
Groups:
- EAS Arm: Subjects who receive a CI and present with a post-operative LFPTA of ≤ 75 dB HL.
  Electric Acoustic Speech Processor: EAS fitting.
  Electric Acoustic Speech Processor: EAS fitting: Electric Acoustic Stimulation for children with post-operative residual low frequency hearing averages of 75 dB HL or better,
Arm/Group | EAS Arm | FES Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 1/16 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EAS Arm (N=16) | FES Arm (N=12)
Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Subject reported a headache and pain with loud sound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03379870/Prot_SAP_000.pdf